CLINICAL TRIAL: NCT03053752
Title: Transcutaneous Electric Nerve Stimulation in Sleep of Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, NADJA MARIA JORGE ASANO, PHD, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAAE: 14877213.8.0000.5208
Record Dates: First submitted 2017-02-08; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcutaneous Electric Stimulation (Experimental): Eight sessions were held, once a week, lasting twenty minutes. For this purpose, the electrodes of the acoustic surface Taichong (LR-3), Hé gǔ (Ll-4), Yanglingquan (GB-34) and Neiguan (PC-6) connected to the TENS equipment (EL 608, brand NKL). The current of choice for a BURST type, with intermittent pulses, isolated at a frequency of 2 Hz, ranging from 1 to 10 mA.
  Interventions: Procedure: Transcutaneous Electric Nerve Stimulation

INTERVENTIONS:
Procedure: Transcutaneous Electric Nerve Stimulation — Eight sessions were held, once a week, lasting twenty minutes. For this purpose, the electrodes of the acoustic surface Taichong (LR-3), Hé gǔ (Ll-4), Yanglingquan (GB-34) and Neiguan (PC-6) connected to the TENS equipment (EL 608, brand NKL). The current of choice for a BURST type, with intermittent pulses, isolated at a frequency of 2 Hz, ranging from 1 to 10 mA.
  Other Names: Tens

SUMMARY:
Sleep disorders are among the non-motor signs more common in Parkinson's disease (PD). This case series evaluated the effects of Transcutaneous Electrical Nerve Stimulation (TENS) on acupoints in the self-assessment of sleep in 14 PD patients classified between stages 1 and 3 of Hoehn and Yahr original (HY). Patients were assessed using the Sleep Scale for Parkinson's Disease (PDSS) and subjected to treatment with eight TENS sessions on acupoints, with the current Burst. We used the paired sample t-test, considering p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic PD between stages 1 and 3 according to the original version of the Hoehn & Yahr (HY) scale

Exclusion Criteria:

* Patients with Mini Mental State Examination (MMSE) lower than 18 points, with other associated neurological diseases and on medication for depression, anxiety, psychosis and sleep inducers.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Scale for Parkinson's disease (PDSS) | 8 weeks
  A self-administered scale designed to assess nighttime sleep problems, sleep disorders and excessive daytime sleep. Consists of 15 items represented by a ruler (10 cm) where the patient indicates the frequency of the symptom from 0 (always)- 10 (never).